CLINICAL TRIAL: NCT06150599
Title: Sacral Neuromodulation for the Treatment of Chronic Pelvic Pain
Brief Title: Sacral Neuromodulation for Chronic Pelvic Pain
Acronym: SNM_CPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Kenneth M Peters, MD, Director and Chair of the Department of Urology, Corewell Health East
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2023-254
Record Dates: First submitted 2023-11-20; First posted 2023-11-29 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pelvic Pain Syndrome
Keywords: Women

STUDY DESIGN:
Intervention Model Description: Single arm and participant-blinded sequential treatment controlled clinical trial. The device will be turned on or off, and settings adjusted at each visit. To minimize bias throughout the study, patients will be blinded to the device settings; however, since there is only one arm, "open label" has been chosen below.
Masking Description: Device is turned on/off, or settings are modified throughout the study. The protocol specifies the exact timing of when the device is turned on/off and or settings are modified. All patients will be on the same schedule. To maintain study integrity, patients will not be informed how device settings are changed; however, since this is a single-arm study, "open label" has been chosen above. During the informed consent process, patients will be explained that throughout the study, the device settings will be modified and that some of these changes may result in symptoms improving while others may cause symptoms to worsen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- SNM for the treatment of CPP (Experimental): Patients will be enrolled based on study eligibility criteria. Eligible patients will be scheduled for a Interstim X implant in the operating room. The procedure is completed under anesthesia, either conscious sedation with intubation or breathing assistance. Under fluoroscopic guidance a standard lead will be introduced. Each electrode on the lead will be tested by confirming motor response on at least 3 of 4 leads. Next the implantable pulse generator will be placed in a subcutaneous pocket and secured. Impedance will be tested, 4 standard programs will be set, and then the device will be shut off. The device settings will be adjusted per protocol and the device will be turned on and off during visits 2-7.
  Interventions: Device: Sacral neuromodulation

INTERVENTIONS:
Device: Sacral neuromodulation — Interstim X, which includes an implantable pulse generator and lead, will be implanted surgically in a single-stage procedure.
  Other Names: SNM; Interstim X

SUMMARY:
Sacral neuromodulation (SNM) is a safe, effective, and minimally invasive FDA approved treatment for urinary and fecal incontinence, urinary frequency, urgency, and urinary retention. In this study we are assessing the effectiveness of sacral neuromodulation in women with suffering from chronic pelvic pain (CPP), through a single device implant procedure.

DETAILED DESCRIPTION:
Despite SNM being available for more than 25 years, there are many things about this technology that remain elusive. Enhancing our understanding of SNM in the chronic pelvic pain (CPP) population can rapidly improve the care of current patients suffering from pelvic pain, as well as help develop future technologies, stimulation paradigms, and lead to effective counseling of patients. CPP is one of most common and challenging conditions for clinicians to treat today. CPP is defined as nonmalignant persistent pain perceived in structures or organs of the pelvis for at least 6 months. As such, CPP can be caused by numerous underlying conditions from gynecological (e.g. endometriosis), gastrointestinal (e.g. celiac disease, irritable bowel syndrome), urological (e.g. interstitial cystitis), musculoskeletal (e.g. fibromyalgia), prostatitis, and neurological/vascular (e.g. spinal cord injury, ilioinguinal nerve entrapment) origin. From a urological perspective, the pain in CPP syndrome can be associated with symptoms suggesting urinary, sexual or bowel dysfunction, and are commonly associated with Overactive Bladder (OAB) symptoms of urinary frequency, urgency, and incontinence. CPP has a debilitating effect on quality of life, leading to other comorbidities such as depression, anxiety, and sleep disorders. CPP is common in both men and women, but occurs more frequently in women. This study will assess the effectiveness of sacral neuromodulation in women.

This is a prospective single arm and single blinded quasi-placebo controlled study. Patients will be blinded to the device settings. For those that qualify, the sacral neuromodulation device will be placed by an experienced physician. After placement in the operating room the device settings will be adjusted. 2 weeks post-operatively participants return and complete study questionnaires. The devices settings will again be adjusted at this visit. The device may turned on/off, or settings modified throughout the study. To maintain study integrity, patients will not be informed how device settings are changed. At each follow up visit, participants will be asked to complete study questionnaires and will have their device settings adjusted. Participants will follow up over a course of 12 months from the time of device implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Female, aged 22-70
4. Chronic pelvic pain (= pain below umbilicus) score of 4 or greater on 10-point VAS, present for 6 months or greater (screening patient)
5. Failed at least 1 or more conservative treatments (e.g. pelvic floor physical therapy, biofeedback, behavioral modification, oral pharmacotherapy, bladder instillations)
6. No changes to current regimen of medications for their pelvic pain for > 4 weeks prior to screening
7. For females of reproductive potential: use of highly effective contraception (e.g. licensed hormonal or barrier methods), for at least 1 month prior to screening and agreement to use such a method during study participation
8. Participant agrees not to start any new treatment interventions for CPP prior to Visit 4 (Primary Endpoint)

Exclusion Criteria:

1. History of any active pelvic cancer
2. Any significant medical condition that is likely to interfere with study procedures, device operation, or likely to confound evaluation of study endpoints
3. Concurrent pain management strategies within the past 3 months that may interfere or mask study intervention (e.g. pelvic floor physical therapy, shockwave therapy, trigger point injections, bladder instillations)
4. Any psychiatric or personality disorder at the discretion of the study physician. This does not include depression or generalized anxiety disorders that are stable.
5. Current symptomatic urinary tract infection (UTI) or more than 6 UTIs in past year
6. Severe or uncontrolled diabetes (A1C > 7, documented in the last 3 months) or diabetes with peripheral nerve involvement
7. Interstitial cystitis diagnosis with Hunner's lesions as this is a severe inflammatory bladder condition that can only be treated with eradication of the lesions or a cystectomy. SNM would be be expected to help for IC with Hunner's lesions
8. Previously implanted with a sacral neuromodulation device or participated in a sacral neuromodulation trial
9. Subject with documented history of allergy to titanium, zirconia, polyurethane, epoxy, or silicone
10. Implantation of spinal cord stimulator and/or drug delivery pumps, whether turned on or off
11. A female who is breastfeeding or of child-bearing potential with a positive urine pregnancy test or not using adequate contraception
12. Current treatment for active malignancy (skin cancers excluded)
13. Patients with spinal pathology that could confound study results. This may include participants with cauda equina syndrome, spinal stenosis, neurogenic claudication, lumbar radiculopathy, patients with primary complaints of leg pain with numbness and or weakness, patients with a primary pain compliant that is vascular in origin, clinical evidence of progressive neurologic pathology, mechanical instability or other spinal pathology that requires surgical intervention, spine or visceral pain secondary to neoplasm, visceral pain in the upper abdomen rather than the pelvis, current diagnosis of fibromyalgia participants with significant cognitive impairment, participants with a condition currently requiring or likely to require use of diathermy or MRI or history of any other condition that in the opinion of the investigator could put the participant at risk or interfere with study results interpretation. (screening patient).
14. Participants involved in ongoing litigation and or injury claims or workers compensation claims.
15. Participation in a current clinical trial or within the preceding 30 days

Note- to preserve the scientific integrity of the study some criteria have been omitted from this posting. All eligibility criteria will be listed at the close of the study.

Ages: 22 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female with female reproductive organs
Enrollment: 25 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
The change in pain score using a 10-point Visual Analogue Scale (VAS) from 2-10 weeks. | Visit 2 (2 weeks post-implant) and Visit 4 (10 weeks post-implant)
  The VAS is a validated tool to determine patient perceived pain. VAS is scored from 0-10, where 0 = no pain and 10 = worst possible pain. The value at Visit 4 (10 weeks post-implant) minus the value at Visit 2 (baseline, 2 weeks post-implant) will be used to calculate change. Negative numbers indicate an improvement in pain, and positive numbers indicate a worsening pain

SECONDARY OUTCOMES:
The change in central sensitization score over 13 months | Visit 2 (2 weeks post-implant) through Visit 8 (an average of 13 months post-implant)
  Change in central sensitization will be assessed using the temporal summation test using the TSA2 AIR system. Temporal summation is considered a manifestation of central sensitization and can be assessed using thermal modalities. It is measured as the magnitude of positive slope of the line fitted to the series of 10 stimuli at the target temperature. A larger slope reflects a higher degree of central sensitization. The central sensitization slope at each treatment visit (visits 3 through 8) minus the slope at visit 2 (baseline, 2 weeks post-implementation) will be recorded and analyzed. A positive number reflects more central sensitization, and a negative number reflects less central sensitization.
Change in pelvic floor pain using a 10-point VAS pain score. | Visit 2 (2 weeks post-implant) through Visit 8 (an average of 13 months post-implant)
  A trained provider will palpate all 4 quadrants of the pelvis, while recording pain scores for each quadrant. The VAS is a validated questionnaire that assesses pain on a scale from 0 = no pain to 10 = worst possible pain. The subject will provide a pain score from 0 - 10 for each of the 4 quadrants assessed. The average pain score of the 4 quadrants is then calculated. The average pain score ranges from 0 to 10. The difference in value from visit 2 (baseline, 2 weeks post implant) minus visit 8 (an average of 13 months post implant) is calculated. A positive number indicates improvement of symptoms. A negative number indicates worsening of symptoms.
Change in severity of overactive bladder symptoms. | Visit 2 (2 weeks post-implant) and Visit 8 (an average of 13 months post-implant)
  The change in OAB symptoms between baseline (visit 2) and subsequent study visits will be assessed using the 6-question Overactive Bladder Questionnaire Short Form (OABq). OABq is a well-established questionnaire used to assess severity of OAB symptoms. The OAB-Q Short Form (SF) consists of two scales assessing symptom bother and health-related quality of life (HR-QOL) in patients with OAB. Each question is rated on a 6 point scale with 1 = Not at all and 6 = A very great deal. Scores can range from 0 to 100, with higher scores indicating more severe symptoms. The change is calculated from the baseline (visit 2, 2 weeks post-implant) minus the value at visit 8 (an average of 13 months post-implant). A positive number indicates improvement of symptoms. A negative number indicates worsening of symptoms.
Change in Female Sexual Function | Visit 2 (2 weeks post-implant) and Visit 8 (an average of 13 months post-implant)
  The Female Sexual Function Index (FSFI) is a 19-question questionnaire evaluating female sexual health in several domains: libido, arousal, lubrication, orgasm, satisfaction, and sexual pain. Each subdomain is scored separately, and the total score calculated. Change in FSFI score will be assessed between baseline (visit 2, 2 weeks-post implant) and visit 8 (an average of 13 months post-implant). A lower FSFI score is equivalent to a higher degree of sexual dysfunction. Scores range from 0 to 36. The change value is calculated from visit 8 (approximately 13 months post-implant) minus visit 2 (baseline, 2 weeks post-implant). A positive number indicates improvement of symptoms. A negative number indicates worsening of symptoms.
Change in mental health and anxiety. | Visit 2 (2 weeks post-implant), Visit 4 (10 weeks post-implant), Visit 5 (an average of 11-15 weeks post-implant), Visit 7 (12 months post-implant), and Visit 8 (an average of 13 months post-implant)
  The Pain Catastrophizing Scale (PCS) is used to determine the impact of SNM on mental health related to pain. Pain catastrophizing is the tendency to describe a pain experience in more exaggerated terms than the average person. The PCS is a validated measure of rumination, magnification, and helplessness related to pain. The PCS has been shown to have adequate to excellent internal consistency. People with higher PCS scores have a tendency to be more likely to report their pain as intense than those with low PCS scores. This objective will be measured at visit 4 (10 weeks post-implant), visit 5 (an average of 11-15 weeks post-implant), visit 7 (12 months post-implant) and visit 8 (an average of 13 months post-implant) and compared to visit 2 scores (baseline, 2 weeks post-implant). Each value will be subtracted from baseline and the difference will be reported. A negative number will indicate more pain catastrophizing, and a positive number will indicate less pain catastrophizing.
Patient satisfaction with sacral neuromodulation treatment | Visit 4 (10 weeks post-implant), Visit 5 (an average of 11-15 weeks post-implant), Visit 7 (12 months post-implant), and Visit 8 (an average of 13 months post-implant)
  Patient satisfaction will be assessed using the Global Response Assessment (GRA) tool on which the patient rates overall patient-perceived symptom improvement on a 7-point scale at visit 4 (10 weeks post-implant) through visit 8 (an average of 13 months post-implant). It is scored as follows: 1 = markedly worse, 2 = moderately worse, 3 = mildly worse, 4 = same (unchanged), 5 = slightly improved, 6 = moderately improved, and 7 = markedly improved. Significant improvement is considered those patient rating their symptoms to be moderately to markedly improved.
Treatment durability measured as change in pain scores from baseline (visit 2) to visit 7 (12 months post-implant) as measured by 10-point visual-analog scale. | Visit 2 (2 weeks post-implant) and Visit 7 (12 months post-implant)
  Treatment durability will be assessed using the 10-point Visual Analogue Scale (VAS) for pain. VAS is scored from 0-10, where 0 = no pain and 10 = worst possible pain. The value at Visit 7 (12 months post-implant) minus the value at Visit 2 (baseline, 2 weeks post-implant) will be used to calculate change. Negative numbers indicate an improvement in pain, and positive numbers indicate a worsening pain
Number of days of carry-over effect after short and long treatment (an average of 13 months post implant) | Visit 8 (an average of 13 months post-implant)
  This objective will be assessed by counting the number of days after visit 7 (12 months post-implant) until the patient reports pain scores that are consistently worsening (prompting the need for an inperson follow-up visit) than reported at visit 2 (baseline, 2 weeks post-implant). This will indicate how long the treatment effect lasts after treatment has been discontinued.
Safety and tolerability: number of adverse events related to the device implantation. | Visit 2 (2 weeks post-implant) through Visit 8 (an average of 13 months post-implant)
  Safety and tolerability of sacral neuromodulation in chronic pelvic pain patients will be assessed by recording the number of adverse events that are determined to be related to device implantation. Adverse events will be assessed at each scheduled study visit or as reported by patients outside study visits.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Corewell Health William Beaumont University Hospital
Locations (1):
- Corewell Health William Beaumont University Hospital, Royal Oak, Michigan, United States